CLINICAL TRIAL: NCT06160531
Title: Randomised, Phase 2a, Double-blind, Placebo-controlled Study to Evaluate the Antiviral Activity Against Influenza Infection, Safety, Tolerability, and Pharmacokinetics of CC-42344 Via a Human Viral Challenge Model in Healthy Participants
Brief Title: Influenza Viral Challenge Study of CC-42344 in Healthy Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cocrystal Pharma, Inc. (Industry)
Collaborators: hVIVO Services Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-42344-P2-001; CPI-CST-001 (Other: hVIVO)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Influenza A
Keywords: Tolerability; Antiviral; Viral challenge model

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CC-42344 Dose 1 (Experimental): Low dose group
  Interventions: Drug: CC-42344
- CC-42344 Dose 2 (Experimental): High dose group
  Interventions: Drug: CC-42344
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-42344 — Anti-influenza A agent
  Arms: CC-42344 Dose 1; CC-42344 Dose 2
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Participants in this study will be given either CC-42344 (one of two dose levels) or placebo orally for 5 days after receiving an influenza (flu) challenge virus. Participants will not know whether they are getting placebo or CC-42344. The amount of virus in nasal samples will be measured over time. Side effects and pharmacokinetics (the amount of CC-42344 in blood) will also be measured.

DETAILED DESCRIPTION:
This is a single-center, phase 2a, randomized, double-blind, placebo-controlled study in healthy adult participants. The primary goal of this study is to assess the antiviral activity of orally administered CC-42344 in an influenza human viral challenge model, and to explore the impact of different dose levels on efficacy. In addition, the safety, tolerability, and pharmacokinetics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Body weight ≥50 kg
* Body mass index ≥18 kg/m2 and ≤35 kg/m2
* Serology results consistent with susceptibility to challenge virus infection

Exclusion Criteria:

* History of or current significant medical condition
* Upper or lower respiratory tract infection within 4 weeks
* Vaccination within 4 weeks

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Area under the influenza viral load-time curve (VL-AUC) of influenza challenge virus | Day 1 to Day 8
  Determined by quantitative real time reverse transcriptase polymerase chain reaction (qRT-PCR) on nasal samples

SECONDARY OUTCOMES:
Maximum viral load | Day 1 to Day 8
  Determined by qRT-PCR on nasal samples
Time to first confirmed nonquantifiable viral assessment | Day 1 to Day 8
  Determined by qRT-PCR on nasal samples
VL-AUC of influenza challenge virus | Day 1 to Day 8
  Determined by viral culture on nasal samples
Maximum viral load | Day 1 to Day 8
  Determined by viral culture on nasal samples
Time to first confirmed nonquantifiable viral assessment | Day 1 to Day 8
  Determined by viral culture on nasal samples
Area under the curve over time of total clinical symptoms score (TSS-AUC) | Day 1 to Day 8
Peak TSS | Day 1 to Day 8
Peak daily symptom score | Day 1 to Day 8
Time to symptom resolution | Day 1 to Day 8
Incidence of adverse events (AEs) | Day 1 to Day 28
  Number of participants with AEs
Incidence of serious adverse events (SAEs) | Day 1 to Day 28
  Number of participants with SAEs
Incidence of AEs related to viral challenge | Day 1 to Day 28
  Number of participants with AEs related to viral challenge
Incidence of SAEs related to viral challenge | Day 1 to Day 28
  Number of participants with SAEs related to viral challenge

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Parker, MMBS, Principal Investigator — hVIVO Services Limited
Locations (1):
- Queen Mary BioEnterprises Innovation Centre, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No